CLINICAL TRIAL: NCT02014220
Title: The Food Intake, Satiety and Blood Glucose After Ingestion of Potato Chips Produced From Three Potato Cultivars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, G. Harvey Anderson, Professor, University of Toronto
Purpose: Prevention
Other Study IDs: Potato study 3: cultivar chips
Record Dates: First submitted 2013-12-08; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Obesity; Overweight; Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Obesity; Overweight; Diabetes Mellitus; Metabolic Syndrome

ARMS (5):
- Atlantic Western chips (Experimental): deep fried potato chips
  Interventions: Other: dietary treatment
- Dakota Pearl chips (Experimental): deep fried potato chips
  Interventions: Other: dietary treatment
- Andover Ontario chips (Experimental): deep fried potato chips
  Interventions: Other: dietary treatment
- white bread with margarine (Experimental): energy control
  Interventions: Other: dietary treatment
- white bread (Experimental): control
  Interventions: Other: dietary treatment

INTERVENTIONS:
Other: dietary treatment

SUMMARY:
Potato is one of the world's most popular foods and is widely accepted as a staple food. The objective of this study is to determine the effect of consuming potato chips from different cultivars on blood glucose, subjective appetite and food intake. It is hypothesized that the chips produced from various potato cultivars will differ in their effect on blood glucose, satiety and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with a body mass index (kg/m2) of 20-24.9

Exclusion Criteria:

* smocking, medication, breakfast skipping, restrained eating

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Dates: Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
blood glucose | 120 min
  Glycaemic response will be measured before the treatment (baseline) and at 15, 30, 45, 60, 90 and 120 min after the treatment. The glucose concentration will be measured in capillary blood using portable glucose meter.

SECONDARY OUTCOMES:
food intake | 120 min
  Ad libidum food intake will be measure at 120 min using test pizza meal. The amount of consumed test meal (g) will be converted to the energy (kcal).

OTHER OUTCOMES:
satiety | 120 min
  Subjective appetite will be measured with visual analogue scales at 0 min immediately before the treatment (baseline) and at 15, 30, 45, 60, 90 and 120 min after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutritional Sciences, Toronto, Ontario, Canada